Web-based Pain Self-Management: Nurse-Guided

NCT03927846

Date: 5/5/2021

Statistical Analysis Plan

| Adjusting for baseline measurement, we used ANCOVA to determine treatment group differences in PROMIS pain intensity and PROMIS pain interference at week 16. |
|---|